CLINICAL TRIAL: NCT00583011
Title: Local Anesthesia and Pain Perception During Amniocentesis: A Randomized Placebo-controlled Trial
Brief Title: Local Anesthesia and Pain Perception During an Amniocentesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AmniocentesisPain
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Pregnancy
Keywords: Amniocentesis; Genetic amniocentesis; Fetal lung maturity; Pain control; Pregnancy; High risk pregnancy
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Local; Amniocentesis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local Anesthesia (Experimental): Local anesthesia group. 2cc of 1% lidocaine with epinephrine administered 2 minutes before amniocentesis, using a 21 gauge needle initially as an intradermal wheal followed by a deeper infiltration of 2cc of 1% lidocaine to the depth of the peritoneum.
  Interventions: Drug: Local Anesthesia
- Placebo-Normal saline (Placebo Comparator): Placebo normal saline group. 2cc of normal saline epinephrine administered 2 minutes before amniocentesis, using a 21 gauge needle initially as an intradermal wheal followed by a deeper infiltration of 2cc of normal saline to the depth of the peritoneum.
  Interventions: Drug: Placebo Group

INTERVENTIONS:
Drug: Local Anesthesia — Local anesthesia: 2 cc of 1% Lidocaine
  Other Names: Amniocentesis
  Arms: Local Anesthesia
Drug: Placebo Group — Placebo Group: 2cc Normal Saline
  Other Names: Amniocentesis
  Arms: Placebo-Normal saline

SUMMARY:
This study is been designed to answer the question of whether local anesthesia (1% lidocaine) decreases the perception of pain associated with amniocentesis in a randomized double blind placebo controlled manner. Our objective is to determine the effect of local anesthesia on the maternal pain perception from an amniocentesis.

DETAILED DESCRIPTION:
Women meeting criteria for project and agreeing to treatment will be randomized into either the 1% Lidocaine or placebo(normal saline) group. The initial injection of either 1% lidocaine or placebo (normal saline) will be administered 2 minutes prior to the amniocentesis procedure. 2cc of 1% lidocaine or placebo (normal saline) will be initially administered as an intradermal "wheal", followed by a deeper infiltration of the 1% lidocaine or placebo (normal saline) to the depth of the peritoneum. All procedures will be performed by either the Maternal-Fetal medicine (MFM) or the reproductive geneticist utilizing continuous ultrasound guidance under sterile conditions. Each woman will be asked to rate their pain perception immediately after the procedure on two pain scales.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* Signed consent to participate in the trial
* Women between the ages of 18 and 45 years
* Gestational ages 15 - 24 weeks

Exclusion Criteria:

* Multiple gestation
* Refusal to participate in the trial
* Known hypersensitivity to lidocaine
* Amniocentesis during this pregnancy
* Amnioinfusion/amnioreduction where the procedure is likely to be prolonged

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2007-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Elimian, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Assessed for eligibility (n=203) Excluded=127(26 not meeting inclusion criteria, 101 declined to participate)
Groups:
- Lidocaine: Local anesthesia group
  Local anesthesia - lidocaine: Local anesthesia: 2 cc of 1% Lidocaine
- Placebo: Placebo normal saline group
  Placebo Group: Placebo Group: 2cc Normal Saline
Period: Overall Study
Arm/Group | Lidocaine | Placebo
Started | 36 | 40
Completed | 36 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lidocaine: Lidocaine group 2cc of 1% lidocaine
- Placebo: Normal saline group 2cc of normal saline
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Placebo | Total
Number analyzed (Participants) | 36 | 40 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 40 | 76
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (6.5) | 30.1 (7.5) | 30.7 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 40 | 76
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 40 | 76

OUTCOME MEASURES:

1. Primary Outcome: Intensity of Perceived Maternal Pain as Measured by the Visual Analogue Scale (VAS)
Description: Visual Analogue Scale (Perpendicular line is drawn at the point that represents pain on a 0-100mm scale, with lower number meaning less pain and the higher number meaning more pain)
Time Frame: Immediately following amniocentesis procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Lidocaine: Lidocaine 2cc of 1% lidocaine group
- Placebo: 2cc of Normal Saline group
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 36 | 40
units on a scale | 9.5 [2.1 to 21.0] | 18.4 [12.9 to 31.3]

2. Secondary Outcome: Intensity of Perceived Maternal Pain as Measured by the 101 Point Numerical Rating Scale (NRS-101)
Description: 101 Point Numerical Rating Scale (NRS-101) (Choose a number that best described pain from 0 to 100 with 0 being least amount of pain and 100 being the worst pain)
Time Frame: Immediately following amniocentesis procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: 2 cc of Normal saline group
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 36 | 40
units on a scale | 15.4 (13.5) | 22.4 (19.8)
Statistical Analysis 1: Comparison: Lidocaine vs Placebo; Test type: Equivalence; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.02

ADVERSE EVENTS:
Time Frame: 6 months
Description: No adverse events
Arm/Group | Lidocaine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/40
Other Adverse Events (participants affected / at risk) | 0/36 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes